CLINICAL TRIAL: NCT02199509
Title: Efficacy of Levetiracetam in Oromandibular and Cranial Dystonia: A Randomized, Double-Blind Placebo-Controlled Cross-Over Study
Brief Title: Efficacy of Levetiracetam in Oromandibular and Cranial Dystonia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 140152; 14-N-0152
Record Dates: First submitted 2014-07-23; First posted 2014-07-24 (Estimated); Results first posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Oromandibular Dystonia; Cranial Dystonia
Keywords: Levetiracetam; Cranial Dystonia; Oromandibular Dystonia
MeSH Terms: interventions — Levetiracetam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Levetiracetam — Anticonvulsant

SUMMARY:
Background:

- People with dystonia cannot control their muscle contractions. This disorder can affect different body areas. When it affects the face, tongue, and jaw, it is called oromandibular dystonia (OMD) or cranial dystonia (CD). Researchers want to find out if a drug that treats seizures may help people with this kind of dystonia.

Objective:

- To see if levetiracetam can improve symptoms of jaw or face dystonia.

Eligibility:

- Adults ages 18 to 80 years with OMD or CD.

Design:

* Participants will be screened with a medical history and physical exam. Researchers will test how severe their dystonia is.
* Participants will have blood drawn through a needle in the arm.
* Participants will be assigned to take either levetiracetam or placebo.
* Phase 1:
* Participants will start with one 500-mg tablet twice daily. The dose will be increased by 500 mg every 3 days. The maximum dose will be 4000 mg a day over 3 weeks. Participants who cannot tolerate that will take the highest dose they can.
* Participants will return for study visits at weeks 3 and 6. They will be asked about their health, side effects, and symptoms of depression. They will have a neurological examination and test of their dystonia.
* After the week 6 visit, participants will taper and stop the study drug over about 1 week.
* Phase 2 begins one week later. Participants will repeat phase 1, but with the other drug.
* After phase 2, participants will return to their usual clinics. They will be told how to stop taking the drug. They will have a follow-up phone call 2 weeks later.

DETAILED DESCRIPTION:
Objectives:

--To determine the efficacy of levetiracetam (LVT) for reducing the symptoms of subjects with oromandibular dystonia (OMD) or cranial dystonia (CD) as assessed by dystonia rating scales and to report all adverse events in this study.

Sample Size and Population:

--We plan to recruit 10 subjects with either primary OMD or CD from the Movement Disorders and Botulinum Toxin (BoNT) Clinics of HMCS.

Design:

--This is a randomized, double-blind placebo controlled cross-over study. All subjects will receive a baseline evaluation and have their dystonia assessed by the eyes, mouth, speech and swallowing subscores of the Burke-Fahn-Marsden (BFM) dystonia scale, and the eyes and upper and lower face, jaw, and tongue subscores of the Global Dystonia Severity (GDS) rating scale. They will then be randomized into two groups. Either LVT or placebo with a titration schedule up to a total daily dose of 4000 mg will be prescribed for six weeks. After week 6, all subjects will undergo tapering and a wash-out period (one week for tapering off and one week for the washout). The two groups will then be switched to the opposite intervention (LVT or placebo), following the same titration and tapering pattern. We will evaluate both groups at weeks 3, 6, 11 and 14 using the same scales. This study requires six outpatient visits to the NIH CC; the total duration of this study will be 15 weeks.

Outcome measurement:

Primary outcome: The percent change of sum of the eyes, mouth, speech and swallowing subscores of BFM dystonia scale at weeks 6 and 14 comparing to the baseline.

Secondary outcome: The percent change of the sum of the eyes, mouth, speech and swallowing subscores of BFM dystonia scale at weeks 3 and 11 and sum of eyes and upper face, lower face and jaw and tongue subscores of the GDS rating scale at weeks 3, 6, 11 and 14 comparing to baseline and all adverse events.

ELIGIBILITY:
* INCLUSION CRITERIA FOR THE PARTICIPANTS:

  1. Be at least 18 years of age and less than or equal to 80 years of age.
  2. Must be able to provide consent.
  3. Primary OMD or CD diagnosed by movement disorders specialist.
  4. No history of receiving LVT.
  5. If the subject is using other medications for their dystonia such as anticholinergics, baclofen, benzodiazepines or tetrabenazine, the dosage must stay the same starting 4 weeks before participation and throughout the duration of the study. Subjects will also be prohibited from starting new medications for their dystonia.
  6. If the subject was injected with BoNT, the latest dose must be injected at least 12 weeks before participation in this study.
  7. Subject is willing to not receive any BoNT injections during the entire study.

EXCLUSION CRITERIA FOR THE PARTICIPANTS:

1. Psychiatric co-morbidities such as depression, psychosis or phobic disorders.
2. Has had a history of brain tumor, stroke, documented history of peripheral trauma to the mouth, jaw or face within a year from the onset of dystonia, epilepsy or seizures.
3. Secondary OMD or CD.
4. Postural instability, frequent falling, severe vertigo or dizziness and severe ataxia.
5. Inability to take medication via oral route due to severe degree of OMD.
6. An estimated creatinine clearance (eCrCL) less than 50 mL/min.
7. Pregnant, lactating or planning to become pregnant in 6 months. Women who are able to get pregnant must be willing to use an effective method of contraception from the time of enrollment until 3 months after the last dose of the study medication.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-07; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hallett, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants between the ages of 18 and 80 with a diagnosis of primary oromandibular or cranial dystonia were recruited from the Movement Disorders and Botulinum Toxin Clinics at the National Institutes of Health and from the Dystonia Global Registry and Dystonia Medical Research Foundation.
Pre-assignment Details: Subjects were excluded if they had a history of depression, psychosis or phobic disorders. One subject was consented but did not participate due to abnormal laboratory finding noted during screening.
Groups:
- Levetiracetam Then Placebo Group: Patients with Primary Oromandibular Dystonia or Cervical Dystonia were given Levetiracetam at maximum tolerated dose for three weeks followed by a Placebo.
- Placebo Then Levetiracetam Group: Patients with Primary Oromandibular Dystonia or Cervical Dystonia were given Placebo for maximum dose for three weeks followed by Levetiracetam.
Period: Overall Study
Arm/Group | Levetiracetam Then Placebo Group | Placebo Then Levetiracetam Group
Started | 3 | 4
Completed | 2 | 3
Not Completed | 1 | 1
Not completed — Suicidal Ideation | 0 | 1
Not completed — Misunderstood titration schedule | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Primary Oromandibular Dystonia or Cranial Dystonia: All participants enrolled in the study.
Arm/Group | Primary Oromandibular Dystonia or Cranial Dystonia
Number analyzed (Participants) | 5
Age, Continuous [Mean (Full Range); unit: years] | 65 [42 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Percent Change of the Sum of the Eyes, Mouth, Speech and Swallowing Subscores of the Burke-Fahn-Marsden (BFM) Dystonia Scale.
Description: The Burke-Fahn-Marsden Dystonia Rating Scale (BFMDRS) is a measure of dystonia severity. The scale consists of evaluation of nine body parts (eyes, mouth, speech, swallowing, neck, trunk, right arm, right leg, left arm and left leg). The severity and provoking factors for each part are rated using a 5-point scale. These range from 0 (indicating no dystonia) to 4 (indicating the presence of dystonia at rest). The primary outcome measure includes the sum of the eyes, mouth, speech and swallowing subscores and represents the percent change from baseline to either 6 weeks or 14 weeks (representing the end of the 3 week period at the maximum tolerated dose for Levetiracetam or Placebo). The total range for these combined sub scores is 0-16, with higher scores indicating more severe dystonia and 0 indicating absence of dystonia.
Time Frame: 6 and 14 weeks compared to baseline
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Levetiracetam Group: Subjects received a starting dose of 500 mg twice daily of levetiracetam. The dose was increased by 250 mg twice daily, every three days until the subject reached a total daily dose of 4000 mg (2000 mg twice daily). The titration took approximately three weeks. At the end of week three, subjects returned to NIH for evaluation. The evaluation included a neurological evaluation using the dystonia rating scales and evaluation of any adverse events including but not limited to depression, hallucination, suicidal ideation or psychosis. Subjects remained on the maximum tolerated dose for three weeks. They returned to NIH at week six for the same evaluation as week three, after which subjects were asked to discontinue the medication in a taper-off fashion over a period of a week and then remain off the medication for another week.
- Placebo Group: Subjects received a starting dose of 500 mg twice daily of placebo. The dose was increased by 250 mg twice daily, every three days until the subject reached a total daily dose of 4000 mg (2000 mg twice daily). The titration took approximately three weeks. At the end of week three, subjects returned to NIH for evaluation. The evaluation included a neurological evaluation using the dystonia rating scales and evaluation of any adverse events including but not limited to depression, hallucination, suicidal ideation or psychosis. Subjects remained on the maximum tolerated dose for three weeks. They returned to NIH at week six for the same evaluation as week three, after which subjects were asked to discontinue the medication in a taper-off fashion over a period of a week and then remain off the medication for another week.
Arm/Group | Levetiracetam Group | Placebo Group
Number analyzed (Participants) | 5 | 5
percent change | 12.16 (29.07) | 31.25 (26.86)

2. Secondary Outcome: Percent Change of the Sum of the Eyes, Mouth, Speech and Swallowing Subscores of Burke-Fahn-Marsten Dystonia Rating Scale (BFM)
Description: The Burke-Fahn-Marsden Dystonia Rating Scale (BFMDRS) is a measure of dystonia severity. The scale consists of evaluation of ten body parts (eyes, mouth, speech, swallowing, neck, trunk, right arm, right leg, left arm and left leg). The severity and provoking factors for each part are rated using a 5-point scale. These range from 0 (indicating no dystonia) to 4 (indicating the presence of dystonia at rest). The secondary outcome measure includes the sum of the eyes, mouth, speech and swallowing subscores and represents the percent change from baseline to either 3 weeks or 11 weeks (representing the end of the three week titration period up to the maximum tolerated dose for Levetiracetam or Placebo). The total range for these combined sub scores is 0-16, with higher scores indicating more severe dystonia and 0 indicating absence of dystonia.
Time Frame: 3 and 11 weeks compared to baseline
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Levetiracetam Group | Placebo Group
Number analyzed (Participants) | 5 | 5
percent change | 14.80 (55.76) | 6.78 (29.37)

3. Secondary Outcome: Percent Change of the Sum of Eyes and Upper Face, Lower Face and Jaw and Tongue Subscores of the GDS Rating Scale
Description: The Global Dystonia Severity Scale provides a severity rating for ten body regions, i.e.,1) eyes and upper face, 2) lower face, 3) jaw and tongue, 4) larynx, 5) neck, 6) shoulder and proximal arm, 7) distal arm and hand including elbow, 8) pelvis and upper leg, 9) distal leg and foot, and 10) trunk. Each body area is rated from 0 to 10, with 0 representing no dystonia present in that body area and 10 representing severe dystonia. The secondary outcome measure includes the sum of the eyes and upper face, lower face and jaw and tongue subscores of the GDS rating scale and represents the percent change from baseline to either 3 and 6 weeks or 11 and 14 weeks (representing the end of the three week titration period (3 weeks and 11 weeks) and the post-3 week period (6 weeks and 14 weeks) at the maximum tolerated dose for Levetiracetam or Placebo). The total range of these combined sub scores is 0-30, with higher scores indicating more severe dystonia and 0 indicating absence of
Time Frame: 3, 6, 11 and 14 compared to baseline
Measure: Mean (Standard Deviation); unit: Percentage of change
Groups:
- Levetiracetam Group at 3 or 11 Weeks; Levetiracetam Group at 6 or 14 Weeks: Subjects received a starting dose of 500 mg twice daily of levetiracetam. The dose was increased by 250 mg twice daily, every three days until the subject reached a total daily dose of 4000 mg (2000 mg twice daily). The titration took approximately three weeks. At the end of week three, subjects returned to NIH for evaluation. The evaluation included a neurological evaluation using the dystonia rating scales and evaluation of any adverse events including but not limited to depression, hallucination, suicidal ideation or psychosis. Subjects remained on the maximum tolerated dose for three weeks. They returned to NIH at week six for the same evaluation as week three, after which subjects were asked to discontinue the medication in a taper-off fashion over a period of a week and then remain off the medication for another week.
- Placebo Group at 3 or 11 Weeks; Placebo Group at 6 or 14 Weeks: Subjects received a starting dose of 500 mg twice daily of placebo. The dose was increased by 250 mg twice daily, every three days until the subject reached a total daily dose of 4000 mg (2000 mg twice daily). The titration took approximately three weeks. At the end of week three, subjects returned to NIH for evaluation. The evaluation included a neurological evaluation using the dystonia rating scales and evaluation of any adverse events including but not limited to depression, hallucination, suicidal ideation or psychosis. Subjects remained on the maximum tolerated dose for three weeks. They returned to NIH at week six for the same evaluation as week three, after which subjects were asked to discontinue the medication in a taper-off fashion over a period of a week and then remain off the medication for another week.
Arm/Group | Levetiracetam Group at 3 or 11 Weeks | Levetiracetam Group at 6 or 14 Weeks | Placebo Group at 3 or 11 Weeks | Placebo Group at 6 or 14 Weeks
Number analyzed (Participants) | 5 | 5 | 5 | 5
Percentage of change | -10.36 (20.06) | 4.11 (32.31) | -16.93 (36.49) | -3.83 (24.80)

ADVERSE EVENTS:
Time Frame: 14 weeks
Groups:
- Levetiracetam: Subjects received a starting dose of 500 mg twice daily of levetiracetam. The dose was increased by 250 mg twice daily, every three days until the subject reached a total daily dose of 4000 mg (2000 mg twice daily). The titration took approximately three weeks. At the end of week three, subjects returned to NIH for evaluation. The evaluation included a neurological evaluation using the dystonia rating scales and evaluation of any adverse events including but not limited to depression, hallucination, suicidal ideation or psychosis. Subjects remained on the maximum tolerated dose for three weeks. They returned to NIH at week six for the same evaluation as week three, after which subjects were asked to discontinue the medication in a taper-off fashion over a period of a week and then remain off the medication for another week.
- Placebo: Subjects received a starting dose of 500 mg twice daily of placebo. The dose was increased by 250 mg twice daily, every three days until the subject reached a total daily dose of 4000 mg (2000 mg twice daily). The titration took approximately three weeks. At the end of week three, subjects returned to NIH for evaluation. The evaluation included a neurological evaluation using the dystonia rating scales and evaluation of any adverse events including but not limited to depression, hallucination, suicidal ideation or psychosis. Subjects remained on the maximum tolerated dose for three weeks. They returned to NIH at week six for the same evaluation as week three, after which subjects were asked to discontinue the medication in a taper-off fashion over a period of a week and then remain off the medication for another week.
Arm/Group | Levetiracetam | Placebo
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levetiracetam (N=5) | Placebo (N=5)
Suicide Ideation (Psychiatric disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes